CLINICAL TRIAL: NCT00825981
Title: Primary and Secondary Hemostasis in Elective Coronary Artery Bypass Graft Surgery
Acronym: HEMOCOR
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Mona Momeni, MD, Cliniques Universitaires saint Luc
Other Study IDs: 2008/10DEC/350
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary artery bypass graft: patients undergoing elective coronary artery bypass graft with or without cardiopulmonary bypass
  Interventions: Other: screening coagulation abnormalities

INTERVENTIONS:
Other: screening coagulation abnormalities — if specific coagulation abnormalities are observed which increase patient's risk of bleeding, appropriate treatment will start

SUMMARY:
Patients undergoing elective coronary artery bypass graft surgery (CABG) are treated with platelet inhibitors to reduce myocardial infarction and mortality.However, this can increase perioperative bleeding. A retrospective analysis of the data in our institution has revealed a significant increase in transfusion requirements after elective CABG since 5 years. The aim of our study is to observe if this increase in transfusion requirements is due to platelet inhibitors or due to other coagulation abnormalities resulting from other anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery bypass graft surgery with or without cardiopulmonary bypass

Exclusion Criteria:

* emergency; redo cardiac surgery; combined cardiac surgery; patients with renal insufficiency; patients with acquired coagulation abnormalities

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: coronary artery bypass graft
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Background] Hertfelder HJ, Bos M, Weber D, Winkler K, Hanfland P, Preusse CJ. Perioperative monitoring of primary and secondary hemostasis in coronary artery bypass grafting. Semin Thromb Hemost. 2005;31(4):426-40. doi: 10.1055/s-2005-916678. PMID 16149021